CLINICAL TRIAL: NCT06876844
Title: Phase II Clinical Study on the Combination of Surufatinib and Envolizumab As Second-line Treatment for Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Surufatinib Combined with Envolizumab As Second-line Treatment for Recurrent/Metastatic HNSCC
Acronym: HNSCC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Guopei Zhu, MD, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMPL-012-SH-HNSCC101
Record Dates: First submitted 2025-02-20; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-12

CONDITIONS: Head and Neck Cancer; Head and Neck Cancer Squamous Cell Carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- combination of Surufatinib and Envolizumab (Experimental): envolizumab: 300 mg subcutaneously every 3 weeks (Q3W); Surufatinib : 200 mg orally within 1 hour after breakfast, once daily continuously every 3 weeks as a treatment cycle until intolerable toxicity or disease progression. If any ≥ Grade 2 treatment-related adverse event occurs during treatment, the dose may be adjusted to 100 mg according to the investigator 's clinical assessment.
  Interventions: Drug: combination of Surufatinib and Envolizumab

INTERVENTIONS:
Drug: combination of Surufatinib and Envolizumab — envolizumab: 300 mg subcutaneously every 3 weeks (Q3W); Surufatinib : 200 mg orally within 1 hour after breakfast, once daily continuously every 3 weeks as a treatment cycle until intolerable toxicity or disease progression. If any ≥ Grade 2 treatment-related adverse event occurs during treatment, the dose may be adjusted to 100 mg according to the investigator 's clinical assessment.

SUMMARY:
This study is a prospective,open-label,single-arm clinical trial to evaluate the efficacy and safety of s Surufatinib combined with envolizumab as second-line treatment of recurrent/metastatic head and neck squamous cell carcinoma .

envolizumab: 300 mg subcutaneously every 3 weeks (Q3W); Surufatinib : 200 mg orally within 1 hour after breakfast, once daily continuously every 3 weeks as a treatment cycle until intolerable toxicity or disease progression. If any ≥ Grade 2 treatment-related adverse event occurs during treatment, the dose may be adjusted to 100 mg according to the investigator 's clinical assessment.

The study is divided into 3 period: Screening, Treatment, and Follow-up. The treatment period is a 3-week treatment cycle. During the treatment period, tumor assessment will be performed by imaging method every 6 weeks (± 7 days) until disease progression (RECIST 1.1) or death (during treatment) or intolerable toxicity. The tumor treatment and survival status after disease progression should be recorded.

Safety measures included: adverse events, laboratory tests, vital signs, and changes in electrocardiogram and cardiac ultrasound.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria for enrollment:

  1. Have fully understood the study and voluntarily signed the informed consent form;
  2. Age: 18-75 years (calculated from the day of informed consent, including the boundary value), both male and female;
  3. Pathologically or histologically confirmed recurrent/metastatic head and neck squamous cell carcinoma (excluding nasopharyngeal carcinoma)
  4. Progressive or recurrent/metastatic disease following first-line systemic therapy within 6 months of completion of concurrent chemoradiation; (first-line systemic therapy includes platinum-based chemotherapy, cetuximab plus chemotherapy, immune checkpoint inhibitors alone or in combination.)
  5. Inability to perform salvage surgery as assessed by oral and maxillofacial surgeons or patient refusal of surgical treatment;
  6. Patients must have at least one measurable lesion (RECIST 1.1);
  7. ECOG performance status 0-2 score;
  8. Expected survival ≥ 6 months;
  9. Vital organs functioning as defined below (no blood components or cell growth factors allowed within 14 days prior to enrollment):
* Absolute neutrophil count ≥ 1.5 x 10 9/L;
* Platelets ≥ 90 × 10 9/L ;
* Hemoglobin ≥ 9 g/dL ;
* Serum albumin ≥ 3 g/dL ;
* Bilirubin ≤ 1.5 times ULN ;
* ALT and AST ≤ 2.5 times ULN ; ( ALT and AST ≤ 5 times ULN if liver metastases );
* Serum creatinine ≤ 1.5 times ULN ; 10. Female patients of childbearing potential voluntarily used highly effective contraception from screening through the designated time after the last dose of study drug (within 1 month after the last dose of Surufatinib or within 2 months after the last dose of envolizumab, whichever came later) and agreed not to donate ovum (oocytes) for reproductive purposes during this period.

All female patients will be considered to be of childbearing potential unless they are naturally postmenopausal, have undergone artificial menopause, or have undergone sterilization (eg, hysterectomy, bilateral adnexectomy, or radiation ovarian irradiation). Male patients with sexual partners of childbearing potential who are willing to use condoms during sex from screening through 3 months after the last dose of study drug and should refrain from donating or freezing sperm during this period.

Exclusion Criteria:

* Any of the following criteria must be excluded from the study plan:

  1. Received previous treatment with Surufatinib and envolizumab, and 6 months with other anti-angiogenic agents;
  2. Received approved or investigational systemic anti-tumor therapy within 4 weeks prior to enrollment, including chemotherapy, radical radiotherapy, biological immunotherapy, targeted therapy;
  3. Participated in other domestic clinical trials of drugs not approved or marketed within 4 weeks before enrollment and received the corresponding investigational drug;
  4. Any major surgery or invasive treatment or operation (except venous catheterization, puncture drainage, etc.) within 4 weeks before enrollment;
  5. International normalized ratio (INR) > 1.5 or activated partial thromboplastin time (APTT) > 1.5 × ULN ;
  6. Clinically significant electrolyte abnormalities as judged by the investigator;
  7. Patients with current hypertension uncontrolled by medications, defined as systolic blood pressure ≥ 140 mmHg and/or diastolic blood pressure ≥ 90 mmHg ;
  8. Patients with currently poorly controlled diabetes (fasting plasma glucose concentration ≥ 10 mmol/L after regular treatment);
  9. Patients with any current disease or condition affecting drug absorption, or patients unable to take oral Surufatinib;
  10. Patients with active gastric and duodenal ulcer, ulcerative colitis and other gastrointestinal diseases or unresected tumors with active bleeding, or other conditions that may cause gastrointestinal bleeding and perforation as judged by the investigator;
  11. Patients with evidence or history of significant bleeding tendency within 3 months prior to enrollment (bleeding > 30 mL with hematemesis, melena, hematochezia within 3 months), hemoptysis (> 5 mL of fresh blood within 4 weeks), or thromboembolic events (including stroke events and/or transient ischemic attack) within 12 months;
  12. Clinically significant cardiovascular disease, including but not limited to acute myocardial infarction, severe/unstable angina pectoris, or coronary artery bypass grafting within 6 months prior to enrollment;
  13. Other malignancies within the last 5 years, except basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix;
  14. Active or uncontrolled serious infection (≥ CTCAE Grade 2 infection);
  15. Known human immunodeficiency virus (HIV) infection; known history of clinically significant liver disease, including viral hepatitis [known hepatitis B (HBV) carriers must exclude active HBV infection, ie, HBV DNA positive (> 1 × 10 4 copies/mL or > 2000 IU/ml); Known hepatitis C virus infection (HCV) and HCV RNA positive (> 1 × 10 3 copies/mL), or other hepatitis, cirrhosis];
  16. Patients with current central nervous system (CNS) metastasis or previous brain metastasis;
  17. Unresolved toxicities above CTCAE Grade 1 due to any prior anticancer therapy, excluding alopecia, lymphopenia, and oxaliplatin-induced neurotoxicity of ≤ Grade 2 ;
  18. Women who are pregnant (positive pregnancy test before medication) or breastfeeding;
  19. Received blood transfusion therapy, blood products and hematopoietic factors such as albumin and granulocyte colony-stimulating factor (G-CSF) within 14 days prior to enrollment;
  20. Tumor involving skin and/or pharyngeal mucosa accompanied by ulceration;
  21. Patients who have a history of psychiatric drug abuse and cannot quit or have mental disorders;
  22. Any other disease, clinically significant metabolic abnormality, physical examination abnormality, or laboratory abnormality that, in the judgment of the investigator, would reasonably suspect that the patient has a disease or condition that would make the use of study drug inappropriate (eg, having a seizure and requiring treatment) or would compromise the interpretation of study results or put the patient at high risk.
  23. Urine routine showed urine protein ≥ 2 + , and 24 hour urine protein > 1.0g ;
  24. Patients with other concomitant diseases that, in the judgment of the investigator, might jeopardize the patient 's safety or might affect the patient' s completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-12-30 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  objective response rate (ORR) (according to RECIST 1.1)

SECONDARY OUTCOMES:
DCR | 1 year
  disease control rate
DOR | 1 year
  duration of response
PFS | 1 year
  progression-free survival
OS | 1 year
  overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No